CLINICAL TRIAL: NCT04262336
Title: Phase 1b Randomized, Double-Blind, Placebo-Controlled, Multicenter Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of Repeated Doses of DB-020 in Patients Receiving Cisplatin
Brief Title: Study to Evaluate Safety and Efficacy of DB-020 to Protect Hearing in Patients Receiving Cisplatin for Cancer Treatment
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Decibel Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: DB-020-002; 1111-1243-8337 (Other: WHO)
Record Dates: First submitted 2020-01-29; First posted 2020-02-10 (Actual); Last update posted 2023-07-06 (Actual); Status verified 2023-07

CONDITIONS: Ototoxicity
Keywords: Ototoxicity; Hearing loss; Chemotherapy-induced
MeSH Terms: conditions — Ototoxicity; Hearing Loss | interventions — sodium thiosulfate; Hyaluronic Acid; Sodium Chloride

STUDY DESIGN:
Intervention Model Description: Part A: DB-020 12% right ear/placebo left ear; DB-020 12% left ear/placebo right ear; DB-020 25% right ear/placebo left ear; DB-020 25% left ear/placebo right ear on Day 1 of every 21 or 28 day cisplatin cycle for up to 6 cycles until cisplatin administration is discontinued
  Part B: DB-020 12% both ears or DB-020-25% both ears on Day 1 of every 21 or 28 day cisplatin cycle for up to 6 cycles until cisplatin administration is discontinued
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double blind
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- DB-020 for Injection, 12%/placebo (Active Comparator): dosage
  Interventions: Drug: DB-020; Drug: Placebo
- DB-020 for Injection, 25%/placebo (Active Comparator): dosage
  Interventions: Drug: DB-020; Drug: Placebo

INTERVENTIONS:
Drug: DB-020 — Injectable sterile viscous solution of DB-020 and sodium hyaluronate in sterile water
  Other Names: Sodium Thiosulfate (STS) pentahydrate formulated in sodium hyaluronate
Drug: Placebo — Injectable sterile viscous solution of sodium hyaluronate in sodium chloride
  Other Names: sodium hyaluronate in sodium chloride

SUMMARY:
The purpose of this study is to evaluate whether DB-020 administered via an injection in the middle ear prevents hearing loss in participants who will receive high doses of cisplatin as part of their treatment for cancer.

DETAILED DESCRIPTION:
Cisplatin is a widely used and effective chemotherapy in the treatment of adult and pediatric solid tumors, including bladder, testicular, head and neck, and lung cancers. Serious side effects of cisplatin treatment include ototoxicity. To date, no approved therapy to prevent or treat ototoxicity exists for people receiving cisplatin treatment, which remains the most common dose-limiting side effect associated with cisplatin administration.

Participants who will be undergoing cancer treatment with high doses of cisplatin every 21 or 28 days will receive IT injection with one ear receiving DB-020 and one ear receiving placebo during each administration. The study will comprise 2 parts. In Part A, eligible participants will be randomized to one of two doses of DB-020. In Part B, participants will be treated with a single dose of DB-020, as selected from data collected in Part A. In both Parts A and B, the ear receiving DB-020 or placebo will be randomized. The choice of dose in Part B will depend on the data from Part A. If appropriate safety and efficacy is observed at either dose level, the Sponsor has the option of dosing at one of these concentrations either unilaterally (ie, with placebo administered in the contralateral ear) or bilaterally (ie, open-label DB-020 administered to both ears) in Part B.

ELIGIBILITY:
Inclusion Criteria:

* Ability to communicate with medical team and staff, willingness to participate in the study, give written informed consent, comply with the study restrictions
* Adults aged 18 years, inclusive, or older
* Treatment for cancer with Intervenous cisplatin once every 21 or 28 days
* Plan to receive a minimum cumulative dose of cisplatin of ≥ 280 mg/m2 over at least three cycles
* Concomitant use of other chemotherapy and radiation is permitted except investigational agents and/or radiation > 35 Grays involving the cochlear area
* Male patients, their female partner(s), and female patients of childbearing potential must agree to use 2 forms of contraception, 1 of which must be a barrier method, during the study and for 90 days after the last study drug administration.
* Male and female patients who consider themselves abstinent, and who agree to remain abstinent during the study and for 90 days after the last study drug administration
* Eastern Cooperative Oncology Group (ECOG) performance status 0 to 2
* Anticipated survival > 1 year
* Normal or not clinically significant otoscopic findings in both ears
* Patient has read, understood, and voluntarily signed the informed consent form.

Exclusion Criteria:

* Female or male patients with female partners who are pregnant, lactating, or planning to attempt to become pregnant during this study or within 90 days after last dose of study drug
* Prior treatment with a cisplatin regimen
* Signs of disturbed integrity of the tympanic membrane on otoscopy or tympanometry
* History of congenital hearing loss
* History of otological surgery (excluding myringotomy tubes or simple tympanoplasty)
* History of sudden hearing loss
* History of conductive hearing loss > 10 decibels at 2 frequencies in either ear
* Diagnosis of Meniere's disease
* Diagnosis of autoimmune middle ear disease
* Hearing loss greater than (not including) 45 decibels Hearing Loss averaged at 6 and 8 kilohertz in either ear
* Asymmetry in hearing thresholds between left and right ear equal to or exceeding 20 decibels at any single frequency or 10 decibels at any 3 consecutive frequencies, up to and including 8 kilohertz
* Previous radiation exposure > 35 Grays to all or part of the cochlea
* Consumption of > 6 grams of salicylate or > 5 grams of acetaminophen (paracetamol) per day for the past month, or aminoglycoside use in the past month
* Use of any investigational drug or device within 30 days prior to the first dose of study medication (6 months for biologic therapies) or 5 half-lives of the investigational drug, if known, whichever time is longer
* History of any significant drug allergy (such as anaphylaxis or hepatotoxicity) and/or allergy to the excipients of the study medications
* Presence of hepatitis C antibody with reflex hepatitis C virus (HCV) RNA testing (if anti-HCV is positive), hepatitis B surface antigen, or HIV antibodies 1 and 2

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2020-02-21 (Actual); Primary Completion 2022-07-30 (Actual); Study Completion 2023-05-23 (Actual)

PRIMARY OUTCOMES:
Number of patients with treatment-emergent Adverse Events (TEAEs) and/or abnormal changes from baseline in clinical laboratory abnormalities and/or vital signs and/or ECG assessments | From screening/baseline (Day -28 to Day -2) or day of first dose of DB-020 (Cycle 1 Day 1) for up to 6 cycles (21 or 28 day cycles) through End of Treatment Visit (28 days after last dose of study drug), up to 196 Days after first dose of study drug
  To investigate the safety and tolerability of DB-020 when given intratympanically to patients receiving cisplatin chemotherapy treatment

SECONDARY OUTCOMES:
Incidence of Ototoxicity measured by American Speech-Language-Hearing Association (ASHA) criteria | Baseline (Day -5 to Day -1) for up to 6 cycles (21 or 28 day cycles) through End of Treatment Visit (28 days after last dose of study drug), up to 196 Days after first dose of study drug
  Air conduction audiometry consists of a set of pure tones presented to the patient through small speakers in a headset, played at carrier frequencies ranging from 250 to 16,000 Hz. Pure tone thresholds are recorded for each frequency tested. Ototoxicity will be defined according to the American Speech-Language-Hearing Association (ASHA) criteria for significant ototoxic change. Significant ototoxic change must meet one of the following three criteria: (i) ≥20 dB decrease at any one test frequency, (ii) ≥10 dB decrease at any two adjacent frequencies, or (iii) loss of response at three consecutive frequencies where responses were previously obtained. The presence of ototoxicity will be calculated for each ear
Changes from Baseline in Pure Tone Threshold Values compared to End of Treatment [Changes in Hearing] | Baseline (Day -5 to Day -1) for up to 6 cycles (21 or 28 day cycles) through End of Treatment Visit (28 days after last dose of study drug), up to 196 Days after first dose of study drug
  Air conduction audiometry consists of a set of pure tones presented to the patient through small speakers in a headset, played at carrier frequencies ranging from 250 to 16,000 Hz. Pure tone thresholds are recorded for each frequency tested. Higher values indicate a greater degree of hearing impairment. Changes from baseline values will be calculated for each frequency and ear as the reported pure tone threshold value minus the baseline value. A negative change from baseline indicates hearing loss
Changes from Baseline in Tinnitus Functional Index (TFI) Total Score compared to End of Treatment [Changes in Hearing] | Baseline (Day -5 to Day -1) for up to 6 cycles (21 or 28 day cycles) through End of Treatment Visit (28 days after last dose of study drug), up to 196 Days after first dose of study drug
  The TFI is a 25-item self-assessment scale comprised of eight subscales (intrusiveness, sense of control, cognitive, sleep, auditory, relaxation, quality of life, and emotional) measuring the impact of tinnitus. Items are scored on a range of 0 to 10. The TFI Total Score is calculated as the mean of the 25 individual item scores multiplied by 10. The Total Score can range from 0 to 100. Higher scores indicate a greater degree of tinnitus-related impairment. Change from baseline values will be calculated as the reported TFI value minus the baseline value. A positive change from baseline indicates more tinnitus-related impairment
Changes from Baseline in Distortion Product Otoacoustic Emission (DPOAE) Values compared to End of Treatment [Changes in Hearing] | Baseline (Day -5 to Day -1) and Cycle 1 Day 1 (21 or 28 day cycles) and End of Treatment Visit (28 days after last dose of study drug), up to 196 Days after first dose of study drug
  Distortion product otoacoustic emission (DPOAE) is defined as sound generated within the cochlea by stimulating the ear with two simultaneous tones of different frequency. DPOAEs serve as an objective measure of hearing sensitivity. Tones will be played from low to high frequencies (1 to 4 kHz) at soft to moderate levels to assess responses at different regions of the inner ear. DP levels will be recorded for each frequency and ear. Higher DP levels indicate more sensitive hearing. Change from baseline values will be calculated as the reported DP level value minus the baseline value. A negative change from baseline indicates less sensitive hearing
Changes from Baseline in Words-in-Noise (WIN) Values compared to End of Treatment [Changes in Hearing] | Baseline (Day -5 to Day -1) and Cycle 1 Day 1 (21 or 28 day cycles) and End of Treatment Visit (28 days after last dose of study drug), up to 196 Days after first dose of study drug
  The WIN test is a series of trials to measure the ability to accurately recognize speech in noise. In each trial, a series of 5 words is read to the listener with the instruction to repeat each word. The number of correct responses is captured. Trials are presented at 7 signal-to-noise ratios, from 0 to 24 dB, in steps of 4 dB. WIN thresholds are then calculated for each ear using the Spearman-Kaerber method. Higher WIN thresholds indicate better word recognition. Change from baseline values will be calculated for each ear as the reported WIN threshold value minus the baseline value. A negative change from baseline indicates worse word recognition
Changes from Baseline in Hearing Handicap Inventory for Adults (HHIA) Total Score compared to End of Treatment [Changes in Hearing] | Baseline (Day -5 to Day -1) and Cycle 1 Day 1 (21 or 28 day cycles) and End of Treatment Visit (28 days after last dose of study drug), up to 196 Days after first dose of study drug
  The Hearing Handicap Inventory for Adults (HHIA) is a 25-item self-assessment scale comprised of two subscales (emotional and social/situational) measuring the impact of hearing loss. Items are scored on a range of 0 to 4. The HHIA Total Score is calculated as the sum of the 25 individual item scores. The HHIA Total Score can range from 0 to 100. Higher scores indicate a greater degree of hearing impairment. Change from baseline values will be calculated as the reported HHIA value minus the baseline value. A positive change from baseline indicates more hearing impairment
Plasma Concentrations of DB-020 | Predose and 0.25 hours prior to cisplatin administration on Cycle 1 Day 1 (21 or 28 day cycles)
Maximum observed plasma concentration (Cmax) of free (unbound) cisplatin | 0.25 hours predose, mid-point of IV infusion, end of infusion, 0.25, 0.5, 1 & 2 hours postdose on Day 1 of each cycle (21 or 28 day cycles)
Area under the plasma concentration-time curve (AUC 0-inf) of free (unbound) cisplatin | 0.25 hours predose, mid-point of IV infusion, end of infusion, 0.25, 0.5, 1 & 2 hours postdose on Day 1 of each cycle (21 or 28 day cycles)
Time to reach maximum observed plasma concentration (tmax) of free (unbound) cisplatin | 0.25 hours predose, mid-point of IV infusion, end of infusion, 0.25, 0.5, 1 & 2 hours postdose on Day 1 of each cycle (21 or 28 day cycles)
Half-life (t1/2) of plasma concentrations of free (unbound) cisplatin | 0.25 hours predose, mid-point of IV infusion, end of infusion, 0.25, 0.5, 1 & 2 hours postdose on Day 1 of each cycle (21 or 28 day cycles)

CONTACTS AND LOCATIONS:
Overall Officials: Pablo LaPuerta, Study Director — Decibel Therapeutics
Locations (8):
- United States (4):
  - University of Miami Health System, Miami, Florida
  - University of Kansas Medical Center, Kansas City, Kansas
  - Northwell Health Cancer Center, Lake Success, New York
  - WVU Cancer Institute, Morgantown, West Virginia
- Australia (4):
  - Queensland Head and Neck Cancer Centre, Woolloongabba, Queensland
  - Peter MacCallum Cancer Centre, Melbourne, Victoria
  - Oncology and Palliative Care Research, Melbourne, Victoria
  - Fiona Stanley Hospital, Clinical Trials Unit Cancer Center, Murdoch, Western Australia

IPD SHARING:
Plan to Share IPD: No